CLINICAL TRIAL: NCT04755452
Title: The Effect of Pneumoperitoneum During Robot Assisted Laparoscopic Renal/ Prostatic Cancer Surgery - a Randomized Clinical Study Investigating Patient and Surgeon Outcome.
Brief Title: The Effect of Pneumoperitoneum (Raised Pressure in the Peritoneal Cavity) During Robotic Kidney/Prostate Cancer Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Hayder Alhusseinawi, Principal investigator, Medical Doctor, PhD student, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: N-2020 00 78
Record Dates: First submitted 2021-02-06; First posted 2021-02-16 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Acute Kidney Injury; Pneumoperitoneum; Kidney
Keywords: Quality of recovery; Surgical rating scale; intra-abdominal pressure; kidney injury biomarkers
MeSH Terms: conditions — Acute Kidney Injury; Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intra-abdominal pressure (Experimental): Intra-abdominal pressure will be set at 7 mm Hg during the procedure.
  Interventions: Procedure: Low intra-abdominal pressure
- High (standard) intra-abdominal pressure (Active Comparator): Intra-abdominal pressure will be set at 12 mm Hg during the procedure.
  Interventions: Procedure: High (standard) intra-abdominal pressure

INTERVENTIONS:
Procedure: Low intra-abdominal pressure — 7 mm Hg pneumoperitoneum during robot-assisted laparoscopic surgery
  Arms: Low Intra-abdominal pressure
Procedure: High (standard) intra-abdominal pressure — 12 mm Hg pneumoperitoneum during robot-assisted laparoscopic surgery
  Arms: High (standard) intra-abdominal pressure

SUMMARY:
Within all the surgical specialties, major surgeries are performed whenever possible, as minimally invasive procedures to reduce blood loss, reduce pain and discomfort after surgery, avoid major scars, provide a faster recovery and thus shorter hospital stay. Such minimally invasive procedures in urinary tract surgeries are often performed as laparoscopic or robotic surgeries where CO2 (carbon dioxide) is insufflated into the abdominal cavity to create a working space for the surgeon's instruments. That high pressure created in the abdominal cavity (pneumoperitoneum) to create a workspace for the surgeon start a series of physiological changes in the heart, lung and kidney.

Today, most laparoscopic, and robotic operations are performed with pneumoperitoneum of approximately 12-15 mm Hg, despite the fact that international guidelines recommend the use of the lowest intra-abdominal pressure (IAP) possible allowing adequate exposure of the operative field rather than using a routine pressure level.

Investigator will conduct a randomized double-blind study involving 120 patients (2 groups of 60). The first group will be operated with standard pressure in the abdominal cavity 12-15 mm Hg (high IAP), patients in the second group will be operated on with a reduced pressure of ≈ 7 mmHg (low IAP).

Investigator would like to assess the practical feasibility of operating under low IAP. Quality of recovery of patients in relation to both physical and mental status, and post-operative use of pain killer will be also investigated using a validated questionnaire . Finally, Invistigator will examine the impact of IAP on post-operative renal function, and risk of kidney injury.

Hypothesis is carrying out laparoscopic/robotic surgeries under low IAP can optimize the post-operative quality of recovery, decrease pain and use of pain killer, improve post-operative renal function, and decrease risk for kidney injury. On the other hand low IAP can risk overview for surgeon, make workspace smaller and raise risk of bleeding.

DETAILED DESCRIPTION:
A total of 120 patients between the ages of 18 and 80 years who were scheduled for elective robotic radical nephrectomy/ prostatectomy will included in the study. This is randomized controlled double-blind clinical trial.

A standard anesthesia protocol will be used in both groups. Bladder catheter inserted by the OP-nurse. After ports installment under IAP of 7 mm Hg, the surgeon leaves the operation field and sits at a surgical console. The ground nurse opens the sealed letter which indicated the pressure for operation (electronic randomization was previously performed by investigator using https://www.graphpad.com/quickcalcs/index.cfm) The required IAP sets by the ground nurse before the surgery started. Assistants are not blinded in the study, but the surgeon is. Intra-abdominal pressure will be maintained at 7 mmHg in Group Low IAP and at 12 mmHg in Group High IAP throughout the surgery. If under operation the surgeon required to raise the IAP because of bad views, or bleeding, he/she can always ask the ground nurse to raise the pressure by 2- or 3-mm Hg at a time until surgeon obtain the preferred view. This involved both groups. Patient will not be excluded from study if pressure increased, but the duration of raised IAP will be registered.

During the operation, the surgical working space will be evaluated by surgeon using an adopted version of SRS (Surgical rating scale). 1st time during mobilization of bowel, 2nd time during renal vascular dissection, and last time when surgeon remove the kidney and set it in the Endobag.

All patients asked to register their 24-hour urine production before the operation day. Intra-operative urine output will be also registered. 10 ml urine will be collected 3 times in order to investigate the risk of Acute Kidney Injury (AKI) by kidney injury biomarker (u-NGAL, og KIM-1). Pre-operatively during urinary catheter placement, 2-hour post-operatively, and 24 hours after operation. Urine samples collected and stored in -80 C for later analyses.

Investigator will test the quality of recovery using a validated Quality of recovery-15 (QoR-15) questionnaire before the surgery and at day 1,3,14,30 post-op.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with kidney/prostate cancer at the department of Urology, Aalborg University Hospital, who are offered radical nephrectomy/prostatectomy.
* Speaks and understands Danish

Exclusion Criteria:

* Patient diagnosed with kidney cancer but can be treated with partial nephrectomy.
* Patients with severe to end stage chronic kidney disease (CKD stage 4-5)
* Inability to understand or comply with instructions.

Withdrawal Criteria:

* Inability to complete the surgery without raising the pneumoperitoneum for low pneumoperitoneum arm.
* Complications that require re-operation which can change the quality of recovery of primary operation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Quality of recovery | fulled by the patient pre-operatively and then on post-operative day 1,3,14 and 30
  Changes in Quality of recovery assessed by QoR-15 Questionaire from pre-operative to day 30 post-operative level. Participiants fill in quistionaire pre-operatively, day 1,3,14,30
Risk Of Acute kidney injury (AKI) | 24 hours after surgery
  post-operative renal function and risk for AKI evaluated by u-NGAL
Surgical rating scale | intra-operative
  assessed 3 times during surgery. 1st during mobilization of bowel, then during renal vessels dissection, and last time during removing and insertion of kidney in the endobag.

SECONDARY OUTCOMES:
post-operative use of painkillers | 24 hours after surgery
  All post-operative painkiller registered and converted to morphine using Morphine Milligram Equivalent (MME)
Intra-operative urine output | intra-operative
Duration of operation in minutes | intra-operative
Intra-operative bleeding in ml | intra-operative
u- KIM-1 level | Before surgery
  Kidney injury molecule in urine
u-NGAL | 24 hours after surgery
  Neutrophil gelatinase-associated lipocalin in urine
u- KIM-1 level | 24 hours after surgery
  Kidney injury molecule in urine
S.creatinine, and eGFR | 24 hours after surgery
  Kidney injury marker
S.creatinine and eGFR | 10 days after surgery
  Kidney injury marker
S.creatinine and eGFR | 21 days after surgery
  Kidney injury marker
Other Kidney injury markers, include; TFF,VEGF, Osteoactivin, Clusterin, and Calbindin | Before surgery
  Kindey injury markers
Other Kidney injury markers, include; TFF,VEGF, Osteoactivin, Clusterin, and Calbindin | 24 hours after surgery
  Kidney injury markers

CONTACTS AND LOCATIONS:
Overall Officials: Hayder Al-husseinawi, M.D., Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg university hospital, Aalborg, North Jutland, Denmark

REFERENCES:
- [Derived] Alhusseinawi H, Sander L, Handberg A, Rasmussen RW, Kingo PS, Jensen JB, Rasmussen S. Impact of low pneumoperitoneum on renal function and acute kidney injury biomarkers during robot-assisted radical prostatectomy (RARP): a randomised clinical trial. J Robot Surg. 2024 Jan 17;18(1):31. doi: 10.1007/s11701-023-01744-2. PMID 38231282
- [Derived] Alhusseinawi H, Sander L, Rosenvinge PM, Jensen SL, Bruun NH, Kingo PS, Jensen JB, Rasmussen S. Low- versus standard- pneumoperitoneum in patients undergoing robot-assisted radical prostatectomy: a randomised, triple-blinded study. BJU Int. 2023 Nov;132(5):560-567. doi: 10.1111/bju.16099. Epub 2023 Jun 26. PMID 37358048